CLINICAL TRIAL: NCT01902979
Title: The Spinal Stenosis Pedometer and Nutrition e-Health Lifestyle Intervention (SSPANLI) Randomized Trial
Brief Title: The Spinal Stenosis Pedometer and Nutrition e-Health Lifestyle Intervention (SSPANLI) Trial
Acronym: SSPANLI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Royal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR290928
Record Dates: First submitted 2013-07-05; First posted 2013-07-18 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Lumbar Spinal Stenosis; Obesity
MeSH Terms: conditions — Spinal Stenosis; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental): In Weeks 1 and 6, people in the intervention group will meet with a Registered Dietitian and an Exercise Physiologist for personalized sessions. They will receive a pedometer and instructions on how to log in to the e-health site (https://sspanli.mtroyal.ca). They will wear the pedometer daily and log in to the website each week for a nutrition education session, a weekly step goal, and tips.
  Interventions: Behavioral: Lifestyle intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle intervention
  Arms: Lifestyle intervention

SUMMARY:
Obesity is one of the most important determinants of quality of life and function. People with lumbar spinal stenosis may be at increased risk of obesity given walking limitations. Spinal stenosis is a very common degenerative condition in people over 45. People with this condition have pain and numbness in the legs during walking, and therefore avoid physical activity. Lack of physical activity is related to weight gain and increased risk of chronic disease. Objective: The objective of this project is test a new e-health (online) pedometer and nutrition intervention aimed at promoting weight loss and increasing physical activity in overweight and obese individuals with spinal stenosis. Methods: The investigators will recruit 88 people with lumbar spinal stenosis who are overweight or obese. Half of these people will receive the 12-week intervention, and the other half will receive usual care (no intervention). In Weeks 1 and 6, people in the intervention group will meet with a Registered Dietitian and an Exercise Physiologist for personalized sessions. They will receive a pedometer and instructions on how to log in to the e-health site (https://sspanli.mtroyal.ca). They will wear the pedometer daily and log in to the website each week for a nutrition education session, a weekly step goal, and tips. The investigators will look to see whether people in the intervention group show greater change in physical activity, body composition and quality of life compared to the individuals who received usual care. Relevance: The increasing number of people with spinal stenosis represents a huge health care burden in Canada. This intervention could provide a new treatment option that would increase mobility, quality of life, and potentially alleviate the need for expensive treatments like surgery. E-health interventions provide an opportunity for patients to take an active role in their own health, and promote behaviour changes that will result in healthier Canadians less likely to access care in the future.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be at least 45 years of age and will have received a diagnosis of lumbar spinal stenosis (LSS) by a spine surgeon who has both examined the patient and reviewed imaging results (MRI or CT). All subjects will be required to have a BMI of 25 kg/m2 or greater (overweight) and to have maintained a stable body weight for the previous 3 months.

Exclusion Criteria:

* any co-morbid conditions that would make participation in a walking program medically inadvisable.
* subjects currently participating in a diet or lifestyle intervention for weight loss or who are on medications known to influence bodyweight or glucoregulation (including antidepressants, sibutramine orlistate, insulin and metformin), will be excluded.

If participants are scheduled for any type of surgery that could impact mobility during the intervention period, they will be removed from the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Percent Fat Mass at 6 months | 6 months
  Fat mass will be assessed at both Baseline and 6 month follow-up using dual energy x-ray absorptiometry and presented as a percentage of total body mass.
Change from Baseline in Mean Number of Steps Per Day at 6 months | 6 months
  Steps per day will be assessed at both Baseline and 6-month follow-up using a pedometer worn for 7 consecutive days
Change from Baseline in Waist Circumference (Centimeters) at 6 months | 6 months
  Waist circumference will be assessed at both Baseline and 6-month follow-up using a tape measure and recorded in centimetres

CONTACTS AND LOCATIONS:
Overall Officials: Christy Tomkins-Lane, Principal Investigator — Mount Royal University
Locations (1):
- Mount Royal University, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Tomkins-Lane CC, Lafave LM, Parnell JA, Krishnamurthy A, Rempel J, Macedo LG, Moriartey S, Stuber KJ, Wilson PM, Hu R, Andreas YM. The spinal stenosis pedometer and nutrition lifestyle intervention (SSPANLI) randomized controlled trial protocol. BMC Musculoskelet Disord. 2013 Nov 14;14:322. doi: 10.1186/1471-2474-14-322. PMID 24228747